CLINICAL TRIAL: NCT05972902
Title: Comparison Between Effects of Dydrogesterone, Cetrorelix Acetate and Triptorelin on Intra Cytoplasmic Sperm Injection Outcomes
Brief Title: Dydrogesterone, Cetrorelix Acetate and Triptorelin in Intra Cytoplasmic Sperm Injection Outcomes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dydrogesterone IVF
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: IVF
Keywords: Dydrogesterone; Intra Cytoplasmic Sperm Injection
MeSH Terms: interventions — Dydrogesterone; cetrorelix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dydrogesterone (Experimental): For pituitary suppression, the patients receives Dydrogesterone (Duphaston 10 mg/twice daily, Abbott Healthcare, America) orally since day 2-3.
  Interventions: Drug: Dydrogesterone
- GnRH antagonist (Active Comparator): For pituitary suppression, the patients receives GnRH antagonist (CETROTIDE 0.25MG , MERCK SERONO, Germany) 0.25 mg/day subcutaneously since the dominant follicles reached the diameter of 12-14 mm till trigger day.
  Interventions: Drug: Cetrorelix acetate
- GnRH agonist (Active Comparator): For pituitary suppression, the patients receives (Decapeptyl, sc 0.1 mg/day) beginning in the afternoon of the 21st day of the cycle prior to stimulation
  Interventions: Drug: Triptorelin

INTERVENTIONS:
Drug: Dydrogesterone — Dydrogesterone molecular structure and pharmacologic effects are closely related to endogenous progesterone
  Other Names: Duphaston
  Arms: Dydrogesterone
Drug: Cetrorelix acetate — GnRH antagonist
  Other Names: cetrotide
  Arms: GnRH antagonist
Drug: Triptorelin — GnRH agonist
  Other Names: Decapeptyl, sc 0.1 mg/day
  Arms: GnRH agonist

SUMMARY:
To compare the effects of Duphaston compared to GnRH agonist and antagonist on the prevention of premature LH surge and quality of retrieved oocytes and embryos in women undergoing intra-cytoplasmic sperm injection.

DETAILED DESCRIPTION:
Study Design:

A randomized clinical trial (RCT).

Study Site:

The study will be conducted at Beni-Suef University Hospital Assisted Reproductive Techniques center. The study population includes all infertile women undergoing IVF at Beni-Suef University ART center will be included. Women will be recruited for enrollment when they come to fertility clinic and scheduled for ICSI trial. They will be counseled and asked to participate in the study after been evaluated to ensure fulfilling inclusion and exclusion criteria.

Study Sample:

The study consisted of 387 women which will be randomized into 3 groups. Women will be enrolled in the study after giving written informed consent. Group (A): 129 Women will start Dydrogesterone group. Group (B): 129 Women will undergo Agonist protocol group. Group (c): 129 Women will undergo Antagonist protocol group.

Study Procedure:

Full history taking. Systematic clinical examination to assess the general condition, body mass index (BMI) and local pelvic physical findings and AFC by trans-vaginal ultrasound on D2 to 3 of menstruation. Routine labs as CBC, liver & kidney functions to exclude general disease as a contraindication for induction or pregnancy. Blood sample obtained for assessment of basal serum levels of FSH, LH, PRL, AMH and E2 on day 3 of the cycle.

Ovarian Stimulation:

#Treatment protocols: The patients begins injections of recombinant FSH (rFSH, Gonal-F; Merck- Serono, Italy) or human menopausal gonadotropin (hp-hMG, Menopur; Ferring Pharmaceuticals, Geneva,Switzerland) since day 2-3 of menstruation, with daily dose of 150-450 IU adjusted according to individual conditions on the basis of the antral follicle count (AFC), age of the woman, body mass index (BMI), and previous ovarian response, according to the standard operating procedures of the center.

For pituitary suppression, the patients received:

* Dydrogesterone (Duphaston 10 mg/twice daily, Abbott Healthcare, America) orally since day 2-3.
* GnRH antagonist (CETROTIDE 0.25MG , MERCK SERONO, Germany) 0.25 mg/day subcutaneously since the dominant follicles reached the diameter of 12-14 mm till trigger day.
* GnRH agonist (Decapeptyl, sc 0.1 mg/day) beginning in the afternoon of the 21st day of the cycle prior to stimulation. The serum LH, estradiol and progesterone levels as well as number and size of follicles will be monitored every 1 to 2 days, starting from stimulation day 5 until the day of hCG injection. The daily dose of rFSH will be adjusted according to patient' s ovarian response, based on serum estradiol levels and the number and size of ovarian follicles as measured by transvaginal ultrasonography.

Triggering and Ovum pick uptake:

Triptorelin (0.2 mg; Decapeptyl, Ferring Pharmaceuticals, the Netherlands) or human chorionic gonadotropin (10000 IU; Choriomon) or Ovitrel 250 mg (Merck Serono, Italy) are given to trigger final maturation of the oocytes. Oocyte retrieval was performed approximately 36 hours later.

Fresh and Frozen Embryo Transfer:

A maximum of 2 embryos will be transferred on day 3 after retrieval under transabdominal ultrasound guidance. Day 3 -5 embryos in the antagonist group and all the viable embryos or blastocysts in the duphaston group are cryopreserved using vitrification.

ELIGIBILITY:
Inclusion Criteria:

* Having indications for ICSI.

Exclusion Criteria:

1. Any known contraindications to the approved fertility drugs.
2. Severe endometriosis.
3. Uterine malformations or abnormal uterine cavity.
4. Uncontrolled endocrinopathies: DM, hyperthyroidism, hypothyroidism.
5. Severe male factor for infertility.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved. | 1cycle (1 month)
  number of oocytes
maturity of oocytes retrieved. | 1 cycle (1month)
  either M2 or M1

SECONDARY OUTCOMES:
Duration of stimulation | 1 ICSI cycle (1 month)
  days till trigger

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided